CLINICAL TRIAL: NCT07067528
Title: The Feasibility and Acceptability of a Diagnostic Algorithm for Timely Post-tuberculosis Lung Disease Diagnosis at Primary Health Care Facilities in Mbarara, Uganda.
Brief Title: The Feasibility and Acceptability of a Post-tuberculosis Lung Disease Diagnostic Algorithm in Uganda.
Acronym: IMPULSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MUST-2025-489; K43TW012781 (NIH)
Record Dates: First submitted 2025-07-03; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Post Pulmonary Tuberculosis; Post-Tuberculous Bronchiectasis
Keywords: tuberculosis; bronchiectasis; fibrosis
MeSH Terms: conditions — Tuberculosis; Bronchiectasis; Fibrosis

STUDY DESIGN:
Intervention Model Description: Pilot cluster randomized trial with four primary health care facilities (clusters) randomized 1:1 to either a structured PTLD diagnostic algorithm (intervention) or usual care (control). Each cluster will contribute an estimated 20 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The diagnostic algorithm arm (Experimental): Primary health care facilities (level three health centers in Uganda) randomized to this arm will implement a diagnostic algorithm developed based on clinical and demographic characteristics earlier in this study to screen tuberculosis (TB) survivors for post-tuberculosis lung disease (PTLD). TB clinicians will use a structured questionnaire and visual aid during routine care to identify PTLD. Patients with suspected PTLD will be referred to Mbarara Regional Referral Hospital, a tertiary center with a functional post-TB care clinic for further evaluation and care
  Interventions: Behavioral: A novel PTLD clinical diagnostic algorithm
- Standard of care arm (No Intervention): Primary health care facilities (level three health centres in Uganda) randomized to this arm will continue routine clinical care after receiving basic training through continuous medical education about post-tuberculosis (TB) lung disease (PTLD) but will not use the diagnostic algorithm. TB clinicians will rely on the guideline-based clinical judgment to identify and refer suspected PTLD cases to Mbarara Regional Referral Hospital.

INTERVENTIONS:
Behavioral: A novel PTLD clinical diagnostic algorithm — A clinical diagnostic algorithm designed to help TB clinicians identify patients at risk of post-tuberculosis lung disease (PTLD) at the end of TB treatment. The algorithm is implemented as a visual aid and structured questionnaire integrated into routine care. Clinicians use it to screen TB survivors and refer suspected PTLD cases to a post-TB clinic for confirmatory evaluation and management.
  Arms: The diagnostic algorithm arm

SUMMARY:
The goal of this clinical trial is to determine whether a structured diagnostic algorithm improves the identification and referral of people with post-tuberculosis lung disease (PTLD) in primary healthcare facilities in Uganda. The clinical trial will, in addition, assess how feasible and acceptable it is for health workers to use this algorithm as part of routine care.

The main trial questions are:

* Does the diagnostic algorithm increase identification and referral of patients with suspected PTLD compared to standard care?
* Is the algorithm feasible to implement and acceptable to health providers and patients in real-world primary health care settings?

The research team will compare four health centre level III (HCIII) facilities ( two using the diagnostic algorithm and two using standard care) to see if the algorithm helps with early diagnosis and referral of PTLD. Health centre level III in Uganda are the primary health facilities and have provision for tuberculosis treatment.

Participants will be screened for PTLD at the time they complete tuberculosis treatment at their local health facility.

At intervention sites, participants will undergo assessment using a structured PTLD diagnostic algorithm developed in earlier stages of this research. The algorithm will be based on a symptom questionnaire and clinical criteria. At control sites, participants will be evaluated using standard practices (consensus clinical definition only).

Participants clinically suspected to have PTLD. will be referred to Mbarara Regional Referral Hospital.

Primary care health facilities will:

* Be randomly assigned to use either the diagnostic algorithm or standard care.
* Receive a baseline training on PTLD and ongoing support through monthly video conference
* Submit triplicate referral forms to track referrals.

DETAILED DESCRIPTION:
Background Tuberculosis (TB) remains a major cause of death globally, with around 1.5 million deaths in 2020. These figures account only for deaths during the active disease phase, not those occurring after microbiologic cure. People who complete pulmonary TB treatment are about four times more likely to die early compared to the general population. Studies show up to 50% of TB survivors report health issues consistent with post-TB lung disease (PTLD). In Malawi, 61% of TB patients still had symptoms at treatment completion, and 28% had irreversible lung damage after five years. Pulmonary TB is now seen as a risk factor for chronic lung disease and poor quality of life. Between 60-90% of TB survivors face limited exercise ability, respiratory symptoms, and reduced quality of life. PTLD is marked by abnormal spirometry (airflow obstruction or low forced vital capacity) and recurrent symptoms often misdiagnosed as TB relapse. This leads to unnecessary TB treatment and drug-related side effects, especially with false-positive Xpert tests in the absence of smear or culture confirmation. PTLD is frequently missed in low-income, TB-endemic settings due to limited resources. Chest imaging shows lung cavities, bronchiectasis, and fibrosis. Spirometry reveals obstructive, restrictive, or mixed patterns, but these tests are not routinely available at primary health centers. Newer tests to distinguish PTLD from TB relapse have not been widely adopted, and culture-the gold standard-is not easily accessible. PTLD receives little attention in global TB guidelines, leading to limited research and diagnostic tools in low- and middle-income countries. Patients at risk of PTLD could be identified using pre-treatment chest X-rays, history, and physical exams, but these approaches are underused. The burden of PTLD varies across sub-Saharan Africa depending on local settings and case definitions. For example, a study in Tanzania found that 90% of people treated for TB in the past five years showed signs of PTLD. Despite a proposed definition from a recent post-TB symposium, no standard PTLD diagnostic criteria exist for low-resource settings. A study in three African countries showed inconsistent PTLD diagnosis, including in Ethiopia, where providers failed to diagnose PTLD in eligible patients. This highlights a critical gap in PTLD diagnosis. More research is needed to create a practical diagnostic tool and understand the barriers to clinical diagnosis. The overall aim of this trial is to build on an existing cohort and design a diagnostic algorithm for PTLD suitable for TB-endemic, low-income settings. PTLD presents a serious but often ignored challenge in TB-endemic areas. People finishing TB treatment should be assessed for overall health, including lung function and nutrition. However, low-income settings lack access to advanced tests like spirometry, relying only on symptom checks. TB programs often overlook PTLD, and health workers at primary facilities may have limited awareness. This trial focuses on improving early PTLD diagnosis at primary health centers, which can impact care for other chronic diseases. While training programs have improved diagnosis of non-communicable diseases, few focus on PTLD. A simple screening algorithm is needed for use at the primary care level. This trial aims to address both personal and system-level barriers to diagnosis. In Uganda, TB treatment is offered at primary health facilities, so early PTLD diagnosis depends on front-line clinicians. PTLD diagnosis is especially difficult at level-three health centers (HC3s) due to limited knowledge, no access to spirometry or imaging, and lack of clear guidelines.

Innovation Innovation A pilot cluster randomized clinical trial in post-TB morbidity is a step closer to improving post-TB care. Importantly, the selected health facilities will focus on post-TB diagnosis and care which has not been part of routine care. Despite the recommendation by the first PTLD symposium, this study aim presents an opportunity to solve this health challenge using locally generated data that can be applied to other low-income settings eliminating a one-size-fits-all approach.

Approach The main idea is that adding a clinical diagnostic algorithm to TB clinicians' workflow will support timely PTLD diagnosis and referrals for advanced care.

Design: This will be a prospective two-arm cluster randomized clinical trial (RCT) using the diagnostic algorithm designed in Aim 1 as the intervention. The primary outcome will be the duration of appropriate referral from level three health centers (HC3s) to a post-TB clinic at Mbarara Regional Referral Hospital (MRRH). The aim is to test the feasibility of implementing a clinical diagnostic algorithm for PTLD aiding clinicians at primary healthcare facilities (HC3s) in making accurate diagnoses of PTLD and facilitating timely referrals for effective treatment.

Study Setting: This study will be conducted at HC3s within Mbarara district Study Participants: The study will involve HC3s selected from the health facilities used for the qualitative interviews in Aim 2. TB clinicians at each health facility will screen individuals who have completed TB treatment for potential PTLD.

Participants: TB clinicians will screen people who completed TB treatment for PTLD.

Procedures: Study Procedures: Four HC3s will be recruited from a catchment area within 10 km radius of MRRH. Facility in-charges identified in Aim 2 will be contacted and requested to participate in the clinical trial. Upon their agreement, the in-charges will sign an informed consent form, following which the facilities will be randomly allocated to either the intervention or control group in a 1:1 ratio. A comprehensive training manual focusing on PTLD aligned with consensus guidelines will be developed for all clinicians at the selected HC3s. This training in form of continuing medical education (CME) will emphasize the significance of PTLD screening in TB survivors presenting with respiratory symptoms after completing TB treatment. The intervention will be the diagnostic algorithm that the investigators developed in Aim 1 as a visual aid whereas the control group will rely their clinical judgment and knowledge gained from the CME. Nurses or clinicians attending to TB patients at each HC3 will be requested to screen for PTLD in all TB survivors declared cured. This includes individuals returning to the TB department of each health facility with symptoms after TB cure. Those with a high suspicion for PTLD based on the diagnostic algorithm (intervention) or clinical judgment (control) will be referred to Mbarara Regional Referral Hospital for further diagnostics and care. A one-page triplicate referral form will be used to track referrals and ensure successful referral completion. The study team will conduct zoom conferences every fortnight with each of the four HC3 teams and to identify registration or referral gaps. No monetary incentives will be provided, but monthly internet and airtime will be provided to the contact health workers involved in the trial. Transport reimbursement and a snack will be provided to patients referred to MRRH. The study will be conducted following the guidelines of good practice in pilot interventional studies. Data Collection: Baseline and endpoint questionnaires will be completed by TB clinicians or any other designated personnel (such as a nurse) in collaboration with our research team. In addition to the routine programmatic TB outcomes documentation, data on patients screened for PTLD will be captured using a standardized data collection tool captured in REDCap. This will include participants demographics and TB treatment history including their prior eCBSS numbers. Facility demographic characteristics will be recorded. The data collection tools will be streamlined to ensure efficient data capture minimizing the potential for questionnaire fatigue. To prevent participants from being recorded at different HC3s due to their close proximity, the investigators will prioritize the recording of eCBSS numbers.

Outcomes: The primary outcome is the time from first visit with PTLD symptoms at HC3 to arrival at MRRH. With no current PTLD screening program, a 50% screening rate will indicate implementation success.

Secondary outcomes:

* Proportion of TB survivors screened for PTLD
* Number of successful referrals to MRRH
* PTLD confirmation rate via imaging/spirometry

Feasibility of a full RCT will be based on:

1. ≥50% facility acceptance rate
2. Completeness of REDCap and algorithm questionnaire data
3. Clinician feedback at study end Data Analysis: Baseline characteristics will be summarized separately for both the intervention and control groups. Feasibility and process evaluation data such as practice recruitment rate and adherence to the intervention will be summarized and presented as percentages. Differences in (1) the primary care interval and (2) screening rate between the two treatment groups will be compared. An exploratory analysis using multivariate regression will be performed to identify factors associated with the ability to implement the intervention

Sample Size: Since this is a feasibility study, study is not powered to test an efficacy hypothesis. However, this study has maximum acceptable confidence interval for an anticipated intra-cluster correlation coefficient of 0.05, at a set cluster size of 20 which is typical for pilot cluster trials, with a coefficient of variation 0.1 and anticipated proportion of 0.5 (50%) for our primary outcome. Therefore FOUR (4) clusters are needed to estimate this proportion (50%) with a lower 0.9 confidence (10% margin of error) limit of 0.27 and upper confidence interval limit 0.73 Key Deliverables: The feasibility of a diagnostic algorithm will be presented in a larger cluster randomized clinical trial to scale up for timely PTLD diagnosis.

Key Deliverable: Demonstrate feasibility of a full-scale cluster RCT to improve PTLD diagnosis.

Challenges and Alternatives: There is a possibility of questionnaire fatigue given the existing programmatic TB questionnaires. However, strategies will be implemented to minimize missing data: Given the average patient load at HC3s TB units (an average 15 patients in a month), our study procedures and short electronic questionnaires are not expected to pose a significant workload. Secondly, monthly airtime and internet will be provided to both groups and an additional incentive such as a mobile phone loan for completing REDCap questionnaires. If the clinical algorithm demonstrated poor diagnostic accuracy, behavioral change will be assessed based on the impact of PTLD-focused CME using the consensus definition as the primary intervention compared to current practice.

ELIGIBILITY:
Inclusion Criteria:

A health facility must meet all of the following criteria to participate in the study.

* Located within a 10 km radius of Mbarara Regional Referral Hospital (MRRH).
* Has an operational TB clinic with at least one designated TB clinician or nurse.
* Facility in-charge (or designated representative) provides written informed consent for participation.
* Willing to implement the PTLD screening procedures and participate in biweekly follow-up communications.
* Agrees to assign a contact staff member to coordinate trial-related activities.

Patients screened at participating facilities must meet all of the following:

* Aged ≥18 years.
* Completed microbiologically confirmed treatment for pulmonary tuberculosis (TB).
* Presenting with persistent or new respiratory symptoms following TB treatment completion.
* Able and willing to provide written informed consent

Exclusion Criteria:

A facility will be excluded if:

* It declines to participate or cannot commit to consistent follow-up activities.
* It lacks the minimum staff or infrastructure to carry out screening and referral procedures.
* It was previously included in a similar PTLD-related intervention trial.

A patient will be excluded if:

* They did complete treatment for pulmonary TB or lack documentation of cure.
* They have a previously confirmed diagnosis of an unrelated chronic respiratory condition (e.g., pulmonary malignancy, cystic fibrosis).
* They were already referred or diagnosed with PTLD prior to this screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Primary care interval | Six months
  The primary care interval (PCI) is the time (in days) between the date a TB survivor presents at a Health Center III (HC3) with symptoms suggestive of post-tuberculosis lung disease (PTLD) and the date they arrive at the post-TB clinic at Mbarara Regional Referral Hospital (MRRH) for confirmatory diagnosis and care. This time will be calculated using patient records and referral logs. The outcome will be compared between the intervention arm (use of diagnostic algorithm) and control arm (standard clinical judgment).

SECONDARY OUTCOMES:
Proportion of TB survivors screened for post-TB lung disease (PTLD) | Six months
  The proportion of TB survivors declared cured who are screened for post-TB lung disease (PTLD) at participating HC3s. This will be presented as a percentage.
Referral completion rate | Six months
  Proportion of TB survivors referred to Mbarara Regional Referral Hospital (MRRH) who successfully arrive at the post-TB clinic for evaluation. This proportion will include all referred patients from participating HC3s
Confirmed post-TB lung disease rate | 6 months
  Proportion of referred patients who receive a confirmed diagnosis of PTLD at Mbarara regional referral hospital post-TB clinic using imaging and/or spirometry.
Screening Fidelity | 6 months
  Implementation fidelity of post-TB lung disease (PTLD) screening, defined as the proportion of eligible TB survivors screened using either the diagnostic algorithm (intervention arm) or clinical judgment (control arm).
Feasibility of data capture | 6 months
  Proportion of eligible TB survivors for whom complete screening and referral data were entered into the REDCap database by health centre-three facility staff.

OTHER OUTCOMES:
Algorithm usability and acceptability | At study termination (6 months)
  Proportion of clinicians in the intervention arm who report that the diagnostic algorithm was easy to use and helpful in clinical decision-making.

CONTACTS AND LOCATIONS:
Locations (1):
- Mbarara University of Science and Technology/Mbarara Regional Referral Hospital, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data leading to published results will be made available upon reasonable request starting 12 months after study completion, for researchers with a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starts 12 months after publication of primary results and will be available for five years
Access Criteria: Scientists, Researchers, patients and organizations that care for lung health will be able to access de-identified participant data. Scientific data generated will be archived in the National Institute of Allergy and Infectious Diseases (NIAID)'s TB Portals Program, a web-based, open-access repository of multi-domain tuberculosis data and tools. TB-Portals program is freely accessible through the Registry of Research Data Repositories. Data will be deposited after the publicaton of our clinical trial results. Our study data will be findable through the NIH data repository. All our publications will be open access and will contain a clause to emphasize that our data is freely and easily accessible through the NIH. The global research community will have access for as long as the data is available at the NIH databases. The NIH data repository will have full control on the decisions about how long to preserve the data.

REFERENCES:
- [Background] Hemming K, Taljaard M, Gkini E, Bishop J. Sample size determination for external pilot cluster randomised trials with binary feasibility outcomes: a tutorial. Pilot Feasibility Stud. 2023 Sep 19;9(1):163. doi: 10.1186/s40814-023-01384-1. PMID 37726817
- [Background] Eldridge SM, Costelloe CE, Kahan BC, Lancaster GA, Kerry SM. How big should the pilot study for my cluster randomised trial be? Stat Methods Med Res. 2016 Jun;25(3):1039-56. doi: 10.1177/0962280215588242. Epub 2015 Jun 12. PMID 26071431
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Uehara S, Hoshi M, Sawada S, Nagatomo T, Ichikawa Y. Monte Carlo calculations of doses to tiles irradiated by 60Co and 252Cf simulating atomic bomb gamma-ray fluences. Health Phys. 1988 Mar;54(3):249-56. doi: 10.1097/00004032-198803000-00001. PMID 3346156
- [Background] Mansell G, Shapley M, Jordan JL, Jordan K. Interventions to reduce primary care delay in cancer referral: a systematic review. Br J Gen Pract. 2011 Dec;61(593):e821-35. doi: 10.3399/bjgp11X613160. PMID 22137419
- [Background] Disbeschl S, Surgey A, Roberts JL, Hendry A, Lewis R, Goulden N, Hoare Z, Williams N, Anthony BF, Edwards RT, Law RJ, Hiscock J, Carson-Stevens A, Neal RD, Wilkinson C. Protocol for a feasibility study incorporating a randomised pilot trial with an embedded process evaluation and feasibility economic analysis of ThinkCancer!: a primary care intervention to expedite cancer diagnosis in Wales. Pilot Feasibility Stud. 2021 Apr 21;7(1):100. doi: 10.1186/s40814-021-00834-y. PMID 33883033
- [Background] Nightingale R, Carlin F, Meghji J, McMullen K, Evans D, van der Zalm MM, Anthony MG, Bittencourt M, Byrne A, du Preez K, Coetzee M, Feris C, Goussard P, Hirasen K, Bouwer J, Hoddinott G, Huaman MA, Inglis-Jassiem G, Ivanova O, Karmadwala F, Schaaf HS, Schoeman I, Seddon JA, Sineke T, Solomons R, Thiart M, van Toorn R, Fujiwara PI, Romanowski K, Marais S, Hesseling AC, Johnston J, Allwood B, Muhwa JC, Mortimer K. Post-TB health and wellbeing. Int J Tuberc Lung Dis. 2023 Apr 1;27(4):248-283. doi: 10.5588/ijtld.22.0514. PMID 37035971
- [Background] Makolkin VI, Petrii VV. [Use of transesophageal electrostimulation of the heart for evaluating the effectiveness of anti-anginal therapy]. Kardiologiia. 1987 Apr;27(4):22-5. Russian. PMID 3599628
- [Background] Willcox PA, Ferguson AD. Chronic obstructive airways disease following treated pulmonary tuberculosis. Respir Med. 1989 May;83(3):195-8. doi: 10.1016/s0954-6111(89)80031-9. PMID 2595036
- [Background] Pexieder T. SEM in studies on abnormal cardiac development. Teratology. 1988 Mar;37(3):289-92. doi: 10.1002/tera.1420370315. No abstract available. PMID 3368882
- [Background] van Kampen SC, Wanner A, Edwards M, Harries AD, Kirenga BJ, Chakaya J, Jones R. International research and guidelines on post-tuberculosis chronic lung disorders: a systematic scoping review. BMJ Glob Health. 2018 Jul 23;3(4):e000745. doi: 10.1136/bmjgh-2018-000745. eCollection 2018. PMID 30057796
- [Background] Khosa C, Bhatt N, Massango I, Azam K, Saathoff E, Bakuli A, Riess F, Ivanova O, Hoelscher M, Rachow A. Development of chronic lung impairment in Mozambican TB patients and associated risks. BMC Pulm Med. 2020 May 7;20(1):127. doi: 10.1186/s12890-020-1167-1. PMID 32381002
- [Background] Meghji J, Mortimer K, Agusti A, Allwood BW, Asher I, Bateman ED, Bissell K, Bolton CE, Bush A, Celli B, Chiang CY, Cruz AA, Dinh-Xuan AT, El Sony A, Fong KM, Fujiwara PI, Gaga M, Garcia-Marcos L, Halpin DMG, Hurst JR, Jayasooriya S, Kumar A, Lopez-Varela MV, Masekela R, Mbatchou Ngahane BH, Montes de Oca M, Pearce N, Reddel HK, Salvi S, Singh SJ, Varghese C, Vogelmeier CF, Walker P, Zar HJ, Marks GB. Improving lung health in low-income and middle-income countries: from challenges to solutions. Lancet. 2021 Mar 6;397(10277):928-940. doi: 10.1016/S0140-6736(21)00458-X. Epub 2021 Feb 22. PMID 33631128
- [Background] Migliori GB, Marx FM, Ambrosino N, Zampogna E, Schaaf HS, van der Zalm MM, Allwood B, Byrne AL, Mortimer K, Wallis RS, Fox GJ, Leung CC, Chakaya JM, Seaworth B, Rachow A, Marais BJ, Furin J, Akkerman OW, Al Yaquobi F, Amaral AFS, Borisov S, Caminero JA, Carvalho ACC, Chesov D, Codecasa LR, Teixeira RC, Dalcolmo MP, Datta S, Dinh-Xuan AT, Duarte R, Evans CA, Garcia-Garcia JM, Gunther G, Hoddinott G, Huddart S, Ivanova O, Laniado-Laborin R, Manga S, Manika K, Mariandyshev A, Mello FCQ, Mpagama SG, Munoz-Torrico M, Nahid P, Ong CWM, Palmero DJ, Piubello A, Pontali E, Silva DR, Singla R, Spanevello A, Tiberi S, Udwadia ZF, Vitacca M, Centis R, D Ambrosio L, Sotgiu G, Lange C, Visca D. Clinical standards for the assessment, management and rehabilitation of post-TB lung disease. Int J Tuberc Lung Dis. 2021 Oct 1;25(10):797-813. doi: 10.5588/ijtld.21.0425. PMID 34615577
- [Background] Singh S, Allwood BW, Chiyaka TL, Kleyhans L, Naidoo CC, Moodley S, Theron G, Segal LN. Immunologic and imaging signatures in post tuberculosis lung disease. Tuberculosis (Edinb). 2022 Sep;136:102244. doi: 10.1016/j.tube.2022.102244. Epub 2022 Aug 11. PMID 36007338
- [Background] Allwood BW, van der Zalm MM, Amaral AFS, Byrne A, Datta S, Egere U, Evans CA, Evans D, Gray DM, Hoddinott G, Ivanova O, Jones R, Makanda G, Marx FM, Meghji J, Mpagama S, Pasipanodya JG, Rachow A, Schoeman I, Shaw J, Stek C, van Kampen S, von Delft D, Walker NF, Wallis RS, Mortimer K. Post-tuberculosis lung health: perspectives from the First International Symposium. Int J Tuberc Lung Dis. 2020 Aug 1;24(8):820-828. doi: 10.5588/ijtld.20.0067. PMID 32912387
- [Background] Sotgiu G, Centis R, Migliori GB. Post-tuberculosis sequelae and their socioeconomic consequences: worth investigating. Lancet Glob Health. 2021 Dec;9(12):e1628-e1629. doi: 10.1016/S2214-109X(21)00454-X. No abstract available. PMID 34798010
- [Background] Binegdie AB, Meme H, El Sony A, Haile T, Osman R, Miheso B, Zurba L, Lesosky M, Balmes J, Burney PJ, Mortimer K, Devereux G. Chronic respiratory disease in adult outpatients in three African countries: a cross-sectional study. Int J Tuberc Lung Dis. 2022 Jan 1;26(1):18-25. doi: 10.5588/ijtld.21.0362. PMID 34969424
- [Background] Byrne AL, Marais BJ, Mitnick CD, Lecca L, Marks GB. Tuberculosis and chronic respiratory disease: a systematic review. Int J Infect Dis. 2015 Mar;32:138-46. doi: 10.1016/j.ijid.2014.12.016. PMID 25809770
- [Background] Nightingale R, Chinoko B, Lesosky M, Rylance SJ, Mnesa B, Banda NPK, Joekes E, Squire SB, Mortimer K, Meghji J, Rylance J. Respiratory symptoms and lung function in patients treated for pulmonary tuberculosis in Malawi: a prospective cohort study. Thorax. 2022 Nov;77(11):1131-1139. doi: 10.1136/thoraxjnl-2021-217190. Epub 2021 Dec 22. PMID 34937802
- [Background] Meghji J, Lesosky M, Joekes E, Banda P, Rylance J, Gordon S, Jacob J, Zonderland H, MacPherson P, Corbett EL, Mortimer K, Squire SB. Patient outcomes associated with post-tuberculosis lung damage in Malawi: a prospective cohort study. Thorax. 2020 Mar;75(3):269-278. doi: 10.1136/thoraxjnl-2019-213808. Epub 2020 Feb 26. PMID 32102951
- [Background] Mbelele PM, Sabiiti W, Heysell SK, Sauli E, Mpolya EA, Mfinanga S, Gillespie SH, Addo KK, Kibiki G, Sloan DJ, Mpagama SG. Use of a molecular bacterial load assay to distinguish between active TB and post-TB lung disease. Int J Tuberc Lung Dis. 2022 Mar 1;26(3):276-278. doi: 10.5588/ijtld.21.0459. No abstract available. PMID 35197168
- [Background] Ravimohan S, Kornfeld H, Weissman D, Bisson GP. Tuberculosis and lung damage: from epidemiology to pathophysiology. Eur Respir Rev. 2018 Feb 28;27(147):170077. doi: 10.1183/16000617.0077-2017. Print 2018 Mar 31. PMID 29491034
- [Background] Pasipanodya JG, Miller TL, Vecino M, Munguia G, Garmon R, Bae S, Drewyer G, Weis SE. Pulmonary impairment after tuberculosis. Chest. 2007 Jun;131(6):1817-24. doi: 10.1378/chest.06-2949. Epub 2007 Mar 30. PMID 17400690
- [Background] Allwood BW, Stolbrink M, Baines N, Louw E, Wademan DT, Lupton-Smith A, Nel S, Maree D, Mpagama S, Osman M, Marx FM, Hoddinott G, Lesosky M, Rylance J, Mortimer K. Persistent chronic respiratory symptoms despite TB cure is poorly correlated with lung function. Int J Tuberc Lung Dis. 2021 Apr 1;25(4):262-270. doi: 10.5588/ijtld.20.0906. PMID 33762069
- [Background] Mpagama SG, Msaji KS, Kaswaga O, Zurba LJ, Mbelele PM, Allwood BW, Ngungwa BS, Kisonga RM, Lesosky M, Rylance J, Mortimer K. The burden and determinants of post-TB lung disease. Int J Tuberc Lung Dis. 2021 Oct 1;25(10):846-853. doi: 10.5588/ijtld.21.0278. PMID 34615582
- [Background] Romanowski K, Baumann B, Basham CA, Ahmad Khan F, Fox GJ, Johnston JC. Long-term all-cause mortality in people treated for tuberculosis: a systematic review and meta-analysis. Lancet Infect Dis. 2019 Oct;19(10):1129-1137. doi: 10.1016/S1473-3099(19)30309-3. Epub 2019 Jul 16. PMID 31324519
- See also: WHO. Global Tuberculosis report — https://www.who.int/publications/i/item/9789240037021

DOCUMENTS (1):
  • Informed Consent Form (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT07067528/ICF_000.pdf